CLINICAL TRIAL: NCT01996228
Title: Reversal of Type 1 Diabetes in Children by Stem Cell Educator Therapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Throne Biotechnologies Inc. (Industry)
Collaborators: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Yong Zhao, MD, PhD, Associate Scientist, Throne Biotechnologies Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0002
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; autoimmune; cord blood stem cell; stem cell educator; immune modulation; children; Control autoimmunity; stimulate the regeneration of islet beta cells
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (1):
- Cord Blood-derived multipotent stem cells (Experimental): Human cord blood-derived multipotent stem cells (CB-SC) display unique phenotypes, such as the expression of embryonic stem (ES) cell markers, multipotential of differentiations, very low immunogenecity, and immune modulations in patients.
  Interventions: Device: Stem Cell Educator

INTERVENTIONS:
Device: Stem Cell Educator
  Other Names: Procedure: Apharesis and Stem Cell Educator Therapy; Biological: Cord blood

SUMMARY:
Type 1 diabetes (T1D) is an autoimmune disease that usually occurs in children and reduces their pancreatic islet beta cells and thereby limits insulin production. Millions of individuals worldwide have T1D, and the number of children with diagnosed or undiagnosed T1D is increasing annually. Insulin supplementation is not a cure. It does not halt the persistent autoimmune response, nor can it reliably prevent devastating complications such as neuronal and cardiovascular diseases, blindness, and kidney failure. A true cure has proven elusive despite intensive research pressure over the past 25 years. Notably, Dr.Zhao and his team have successfully developed a groundbreaking technology Stem Cell Educator therapy (Zhao Y, et al.BMC Medicine 2011, 2012). To date, clinical trials in adult patients have demonstrated the safety and efficacy of Stem Cell Educator therapy for the treatment of T1D and other autoimmune-associated diseases. Here, the investigators will evaluate the safety and efficacy of Stem Cell Educator therapy in children with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 1. T1D patients are screened for enrollment in the study if both clinical signs and laboratory tests meet the diagnosis standards of American Diabetes Association.

  2. Children from 3 through 18 years old and body weight > 15 kg.

  3. Presence of at least one autoantibody to the pancreatic islet β cells (IA-2, GAD, ICA, ZnT8, or IAA).

  4. Written informed consent from the child and child's parents or legal representative.

Exclusion Criteria:

* 1. Any clinically significant diseases in liver, kidney, and heart.

  2. Additional exclusion criteria include no immunosuppressive medication, no viral diseases or diseases associated with immunodeficiency

  3. Significantly abnormal hematology results at screening.

  4. Presence of any infection diseases or inflammation conditions, including active skin infections, flu, fever, upper or lower respiratory track infections.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2013-11; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Autoimmune control | 90 days post treatment
  Before treatment, test autoimmune-related markers as baseline; After treatment for 90 days, repeat testing autoimmune-related markers.

SECONDARY OUTCOMES:
Metabolic control | 3-24 months post treatment
  Before treatment, test for C-peptide levels and HbA1C as baseline; After treatment, test C-peptide levels and HbA1C on the 3rd month.
  1. Analysis of islet beta cell function
  2. Test for C-peptide levels on every 6 month;
  3. Full evaluation of islet beta cell function after two years.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Zhao, MD,PhD, Study Chair — Tianhe Stem Cell Biotechnologies; Zhiguang Zhou, Md,PhD, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (1):
- The Second Xiangya Hospital, Changsha, Hunan, China

REFERENCES:
- [Background] Zhao Y, Jiang Z, Zhao T, Ye M, Hu C, Yin Z, Li H, Zhang Y, Diao Y, Li Y, Chen Y, Sun X, Fisk MB, Skidgel R, Holterman M, Prabhakar B, Mazzone T. Reversal of type 1 diabetes via islet beta cell regeneration following immune modulation by cord blood-derived multipotent stem cells. BMC Med. 2012 Jan 10;10:3. doi: 10.1186/1741-7015-10-3. PMID 22233865
- [Background] Zhao Y, Jiang Z, Zhao T, Ye M, Hu C, Zhou H, Yin Z, Chen Y, Zhang Y, Wang S, Shen J, Thaker H, Jain S, Li Y, Diao Y, Chen Y, Sun X, Fisk MB, Li H. Targeting insulin resistance in type 2 diabetes via immune modulation of cord blood-derived multipotent stem cells (CB-SCs) in stem cell educator therapy: phase I/II clinical trial. BMC Med. 2013 Jul 9;11:160. doi: 10.1186/1741-7015-11-160. PMID 23837842
- [Background] Zhao Y. Stem cell educator therapy and induction of immune balance. Curr Diab Rep. 2012 Oct;12(5):517-23. doi: 10.1007/s11892-012-0308-1. PMID 22833322
- [Background] Zhao Y, Mazzone T. Human cord blood stem cells and the journey to a cure for type 1 diabetes. Autoimmun Rev. 2010 Dec;10(2):103-7. doi: 10.1016/j.autrev.2010.08.011. Epub 2010 Aug 20. PMID 20728583
- See also: Tianhe Stem Cell Biotechnologies — http://www.tianhecell.com